CLINICAL TRIAL: NCT06359301
Title: An Open Label, Observational, Prospective, Longitudinal Cohort Study to Evaluate Safety, Clinical and Radiographic Outcomes of Total Hip Arthroplasty With DELTA Revision Cup
Brief Title: H-34 DELTA Revision Cup
Status: Recruiting | Type: Observational
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Other Study IDs: H-34
Record Dates: First submitted 2024-03-15; First posted 2024-04-11 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Hip, Osteoarthritis
Keywords: revision
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: DELTA Revision acetabular cup — Total hip arthroplasty

SUMMARY:
THis study is aimed to provide a clinical and radiographic evaluation of 49 suitable subjects who underwent a total hip arthroplasty with DELTA Revision acetabular cup.

DETAILED DESCRIPTION:
This is an observational study designed to reflect real life clinical practice as closely as possible. Thus, clinicians are free to choose the method to implant and total hip arthroplasty in accordance with the current local Delta Revision acetabular cup Indication for Use and current clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* male or female in whom a decision has already been made to perform a total hip arthroplasty with DELTA Revision acetabular cup as per indication for use. The decision to implant DELTA revision acetabular cup must be taken prior to, and independently from the decision to enroll the patient. This decision should be made in accorsance with routine clinical practice at the study site concerned.
* Age ≥ 18 years old
* All patients mist give written informed consent approved by the study site's Institutinal Review Board (IRB)/Ethical Committee (EC)
* Patient is able to comply with the protocol

Exclusion Criteria:

* Adult patients with any DELTA Revision acetabular cup contraindication for use as reported in the current local instruction for use.
* For female patiens, current pregnancy and/or lactation or planning a pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of 49 consecutive subjects who underwent a THA with the DELTA Revision acetabular cup at the Independent Public Clinical Hospital Prof. Adama Grucy CMKP.
  Subjects who do not meet all the inclusion criteria or meet any exclusion criteria are excluded from study participation and should be considered as a Screening Failure.
  Subjects who meet all the inclusion criteria and none of the exclusion criteria and agree to participate in the study signing the Informed Consent Form are enrolled.
Sampling Method: Probability Sample
Enrollment: 49 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Harris Hip Score (HHS) | From preoperative to 2 years after surgery
  Overall score from 0 to 100, with 100 being the best outcome

SECONDARY OUTCOMES:
ROM measurement | From preoperative to 2 years after surgery
  Functional changes in ROM measurements from pre-operative (baseline), discharge, 2 months, 6 months, 1 year and 2 years
Oxforn Hip Score (OHS) | From preoperative to 2 years after surgery
  Overall score from 0 to 48, with 48 being the best outcome
Survival rate | 2 years
  Survival rate expressed with Kaplan-Meier estimator at 2 years after surgery
Radiographic implant evaluation and stability assessment of the DELTA Revision acetabular cup | From preoperative to 2 years after surgery
  The treated hip is analyzed postoperatively based on anteroposterior and lateral x-rays view of the knee to check for radiographic stability and radiographically detectable complications
Incidence, type and severity of all the Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Device Effects (ADEs), and Serious Adverse Device Effects (SADEs) occurred at each follow-up | From preoperative to 2 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jerzy Bialecki, Principal Investigator — Samodzielny Publiczny Szpital Kliniczny im. Prof. Adama Grucy CMKP
Locations (1):
- Samodzielny Publiczny Szpital Kliniczny im. Prof. Adama Grucy CMKP, Otwock, Poland

IPD SHARING:
Plan to Share IPD: No